CLINICAL TRIAL: NCT03270449
Title: A Multi-disciplinary, Community-based Group Intervention for Fibromyalgia: A Pilot Randomized Controlled Trial
Brief Title: Community-based Intervention for Fibromyalgia: A Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Rheumatology Association (Other); Interior Health (Industry)
Responsible Party: Principal Investigator, Nelly Oelke, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H17-01782
Record Dates: First submitted 2017-08-21; First posted 2017-09-01 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; community-based; multidisciplinary
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary intervention (Experimental): The 10-week intervention will include twice weekly 1-2 hours sessions with multiple professional team members to undergo education and exercise sessions. The multidisciplinary team will consist of a rheumatologist, rheumatology nurse, dietitian, physiotherapist, a trained exercise therapist, a physiologist who specializes in pain management, a psychiatrist and a mental health clinician. All intervention team members have expertise in working with individuals with chronic pain conditions. General disease information, current best practices and techniques such as self-pain management, pacing, sleep hygiene, approach to a healthy lifestyle and weight loss will be discussed. The total number of hours for the 10 week intervention is 31 hours.
  Interventions: Other: Multidisciplinary intervention
- Usual care (No Intervention): Usual care involves being referred to the local rheumatologist involved in the study. The rheumatologist and the rheumatology nurse will see the control group patients during a one hour one on one consultation appointment. During that time the patient's history will be taken, physical exam performed and investigations analyzed. If a diagnosis of fibromyalgia is confirmed, the rheumatologist and nurse will counsel the patient and provide resources for self directed management. Unless there is a concern of an alternative diagnosis, follow up will not be arranged.

INTERVENTIONS:
Other: Multidisciplinary intervention — 10 week multidisciplinary education and exercise
  Arms: Multidisciplinary intervention

SUMMARY:
Fibromyalgia (FM) is a multi-factorial chronic pain condition characterized by fluctuating and heterogeneous symptoms. This leads to both reduced patient function and quality of life and consequentially, significant economic burden on the society. Although numerous pharmaceutical and multi-treatment approaches exist, there is lack of an integrated multidisciplinary model of care for these patients. Such a system is hypothesized to be beneficial for the patients and would help them regain function and significantly improve their quality of life. The primary aim of this pilot clinical trial is to evaluate the effectiveness of an integrated community-based multidisciplinary model of care for FM patients in Penticton and surrounding areas. The comprehensive 10 week intervention will provide care from a team of health care providers (psychiatrist, physiotherapist, certified exercise therapist, dietitian, rheumatologist, and mental health clinician). Patients will also attend a peer led pain self-management support group provided by the Arthritis Society. The study aims at educating these patients about self-management of their symptoms such as chronic pain, weight, sleep and mood disorders. The integration of health care between the different providers will be achieved by "huddle" sessions that will be conducted on a monthly basis. The evaluation of the study outcomes will be based on the RE-AIM framework. Data will be collected through patient questionnaires, healthcare utilization data, and interviews with providers. Data analysis will involve thematic analysis of qualitative data and statistical methods for quantitative data.

ELIGIBILITY:
Inclusion Criteria:

* formal diagnosis of FM
* resident of Penticton or surrounding area
* adults, aged 19 and older
* fluent in English or bring a family member/friend to assist with translation
* capacity to provide informed consent

Exclusion Criteria:

* patients with a severe and/or chronic medical or psychiatric condition that would impact ability to participate in the intervention
* patients who are pregnant or lactating

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Patient-perceived quality of care | Change from baseline in perceived quality of care at 10 weeks and 6 months
  Patient assessment of care received as measured by the Patient Assessment of Chronic Illness Care Questionnaire

SECONDARY OUTCOMES:
Daily function #1 | Change from baseline in daily function at 10 weeks and 6 months
  Physical disease and mental health related functioning as measured by Revised-Fibromyalgia Impact Questionnaire
Daily function #2 | Change from baseline in daily function at 10 weeks and 6 months
  Mental health related functioning as measured by Hospital Anxiety and Depression scale
Health care utilization (physician visits) | Change from baseline in physician visits at 6 months
  Number of physician visits
Health care utilization (emergency visits) | Change from baseline in emergency department visits at 6 months
  Number of emergency department visits

OTHER OUTCOMES:
Sleep quality | Change from baseline in sleep quality at 10 weeks
  Quality of sleep as measured by Sleep scale - medical outcome scale
Sleep quality | Change from baseline in sleep quality at 6 months
  Quality of sleep as measured by Sleep scale - medical outcome scale
Attitudes of pain | Change from baseline in pain attitudes at 10 weeks and 6 months
  Measurement of pain through Survey of brief attitudes of pain
Irritability | Change from baseline in irritability at 10 weeks
  Irritability measured by Brief Irritability Test (BITe) questionnaire
Irritability | Change from baseline in irritability at 6 months
  Irritability measured by Brief Irritability Test (BITe) questionnaire
Patient perspectives on self-management resources | 10 weeks
  Questionnaire to be administered to gather patient perspectives on self-management resources offered via hard copy, online, and social media
Patient perspectives on self-management resources | 6 months
  Questionnaire to be administered to gather patient perspectives on self-management resources offered via hard copy, online, and social media
Provider perspectives on quality of care | 18 months
  Interviews will be conducted to gather providers' perspectives on the model of care

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Teo, Principal Investigator — University of British Columbia
Locations (1):
- Balfour Medical Centre, Penticton, British Columbia, Canada

REFERENCES:
- [Background] Fitzcharles MA, Ste-Marie PA, Goldenberg DL, Pereira JX, Abbey S, Choiniere M, Ko G, Moulin DE, Panopalis P, Proulx J, Shir Y; National Fibromyalgia Guideline Advisory Panel. 2012 Canadian Guidelines for the diagnosis and management of fibromyalgia syndrome: executive summary. Pain Res Manag. 2013 May-Jun;18(3):119-26. doi: 10.1155/2013/918216. PMID 23748251
- [Background] Schaefer C, Chandran A, Hufstader M, Baik R, McNett M, Goldenberg D, Gerwin R, Zlateva G. The comparative burden of mild, moderate and severe fibromyalgia: results from a cross-sectional survey in the United States. Health Qual Life Outcomes. 2011 Aug 22;9:71. doi: 10.1186/1477-7525-9-71. PMID 21859448
- [Background] Lachaine J, Beauchemin C, Landry PA. Clinical and economic characteristics of patients with fibromyalgia syndrome. Clin J Pain. 2010 May;26(4):284-90. doi: 10.1097/AJP.0b013e3181cf599f. PMID 20393262
- [Background] Thompson JM, Luedtke CA, Oh TH, Shah ND, Long KH, King S, Branda M, Swanson R. Direct medical costs in patients with fibromyalgia: Cost of illness and impact of a brief multidisciplinary treatment program. Am J Phys Med Rehabil. 2011 Jan;90(1):40-6. doi: 10.1097/PHM.0b013e3181fc7ff3. PMID 20975520
- [Background] Winkelmann A, Perrot S, Schaefer C, Ryan K, Chandran A, Sadosky A, Zlateva G. Impact of fibromyalgia severity on health economic costs: results from a European cross-sectional study. Appl Health Econ Health Policy. 2011 Mar 1;9(2):125-36. doi: 10.2165/11535250-000000000-00000. PMID 21332254
- [Background] Bellato E, Marini E, Castoldi F, Barbasetti N, Mattei L, Bonasia DE, Blonna D. Fibromyalgia syndrome: etiology, pathogenesis, diagnosis, and treatment. Pain Res Treat. 2012;2012:426130. doi: 10.1155/2012/426130. Epub 2012 Nov 4. PMID 23213512
- [Background] Gaglio B, Shoup JA, Glasgow RE. The RE-AIM framework: a systematic review of use over time. Am J Public Health. 2013 Jun;103(6):e38-46. doi: 10.2105/AJPH.2013.301299. Epub 2013 Apr 18. PMID 23597377
- [Background] Richards L, Morse J. Read me first for a users guide to qualitative methods. (3rd ed.) Sage Publications, Inc. 2013.
- [Background] Verbeke G, Molenberghs G. Linear mixed models for longitudinal data. Springer Science & Business Media; 2009.
- [Background] Glasgow RE, Wagner EH, Schaefer J, Mahoney LD, Reid RJ, Greene SM. Development and validation of the Patient Assessment of Chronic Illness Care (PACIC). Med Care. 2005 May;43(5):436-44. doi: 10.1097/01.mlr.0000160375.47920.8c. PMID 15838407
- [Background] Bennett RM, Friend R, Jones KD, Ward R, Han BK, Ross RL. The Revised Fibromyalgia Impact Questionnaire (FIQR): validation and psychometric properties. Arthritis Res Ther. 2009;11(4):R120. doi: 10.1186/ar2783. Epub 2009 Aug 10. PMID 19664287
- [Background] Nam S, Tin D, Bain L, Thorne JC, Ginsburg L. Clinical utility of the Hospital Anxiety and Depression Scale (HADS) for an outpatient fibromyalgia education program. Clin Rheumatol. 2014 May;33(5):685-92. doi: 10.1007/s10067-013-2377-1. Epub 2013 Sep 1. PMID 23995734
- [Background] Cappelleri JC, Bushmakin AG, McDermott AM, Dukes E, Sadosky A, Petrie CD, Martin S. Measurement properties of the Medical Outcomes Study Sleep Scale in patients with fibromyalgia. Sleep Med. 2009 Aug;10(7):766-70. doi: 10.1016/j.sleep.2008.09.004. Epub 2009 Jan 29. PMID 19185539
- [Background] Tait RC, Chibnall JT. Development of a brief version of the Survey of Pain Attitudes. Pain. 1997 Apr;70(2-3):229-35. doi: 10.1016/s0304-3959(97)03330-7. PMID 9150298